CLINICAL TRIAL: NCT03451292
Title: Prevention of Mortality With Long-Term Administration of Human Albumin in Subjects With Decompensated Cirrhosis and Ascites
Brief Title: Effects of Long-Term Administration of Human Albumin in Participants With Decompensated Cirrhosis and Ascites
Acronym: PRECIOSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Collaborators: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IG1601; 2016-001789-28 (EudraCT Number)
Record Dates: First submitted 2018-02-12; First posted 2018-03-01 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Decompensated Cirrhosis and Ascites
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SMT + Albutein 20% (Experimental): Participants received Albutein 20%, at a dose of 1.5 grams/kilograms (g/kg), based on their body weight (maximum 100 grams per participant), as an intravenous (IV) infusion on Day 1, followed by the same dose of Albutein 20% every 10±2 days along with standard medical treatment (SMT) administered as per institution standards for the management of decompensated cirrhosis up to 12 months.
  Interventions: Drug: Albutein 20%; Other: SMT
- SMT (Active Comparator): Participants received SMT up to 12 months as per institution standards for the management of decompensated cirrhosis.
  Interventions: Other: SMT

INTERVENTIONS:
Drug: Albutein 20% — Injectable solution
  Arms: SMT + Albutein 20%
Other: SMT — Participants received SMT according to institution standards for the management of decompensated cirrhosis.

SUMMARY:
This is a phase 3, multicenter, randomized, controlled, parallel-group, and open-label clinical study to evaluate the efficacy of standard medical treatment (SMT) + Albutein 20% administration versus SMT alone in participants with decompensated cirrhosis and ascites. The study population will consist of participants being discharged after hospitalization for acute decompensation of liver cirrhosis with ascites (or with prior history of ascites requiring diuretic therapy) with or without acute-on-chronic liver failure (ACLF) at admission or during hospitalization but without ACLF at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥18 years of age.
* Participants with diagnosis of liver cirrhosis (based on clinical, laboratory, endoscopic, and ultrasonographic features or on histology).
* Participants who have been hospitalized for acute decompensation of liver cirrhosis with ascites (or with prior history of ascites requiring diuretic therapy) with or without ACLF at admission or during hospitalization but without ACLF at Screening.
* In participants with cirrhosis due to hepatitis B virus, decompensation must occur in the setting of continuous (no less than 3 months) appropriate antiviral therapy.
* In participants with cirrhosis due to hepatitis C virus, only decompensated participants who will not receive antiviral therapy during the study period will be included (Participants receiving antiviral therapy within 14 days prior to enrollment cannot be included in the study).
* In participants with cirrhosis due to autoimmune hepatitis, decompensation must occur in the setting of continuous immunosuppressive therapy.
* Participants must be willing and able to provide written informed consent or have an authorized representative able to provide written informed consent on behalf of the participant in accordance with local law and institutional policy.
* Chronic liver failure-consortium acute decompensation (CLIF-C AD) score > 50 points at screening.

Exclusion Criteria:

* Participants with ACLF at Screening
* Participants with type 1 hepatorenal syndrome (HRS) currently on treatment with vasoconstrictors or hemodialysis.
* Participants with transjugular intrahepatic portosystemic shunt (TIPS) or other surgical porto-caval shunts.
* Participants with refractory ascites as defined by the International Club of Ascites (ICA) criteria without any other event of acute decompensation.
* Participants receiving dual anti-platelet therapy or anti-coagulant therapy (exception: deep vein thrombosis (DVT) prophylaxis).
* Participants with ongoing endoscopic eradication of esophageal varices with ≤ 2 endoscopic sessions completed before screening.
* Participants with evidence of current locally advanced or metastatic malignancy.
* Participants with acute or chronic heart failure (New York Heart Association [NYHA]).
* Participants with severe (grade III or IV) pulmonary disease (Global Obstructive Lung Disease [GOLD]).
* Participants with nephropathy with renal failure with serum creatinine >2 milligrams/deciliters (mg/dL) or systemic hypertension.
* Participants with severe psychiatric disorders.
* Participants with a known infection with human immunodeficiency virus (HIV) or have clinical signs and symptoms consistent with current HIV infection.
* Females who are pregnant, breastfeeding, or if of childbearing potential, unwilling to practice effective methods of contraception
* Participants with previous liver transplantation.
* Participants with known or suspected hypersensitivity to albumin.
* Participants participating in another clinical study within 3 months prior to screening.
* Participants with active drug addiction (exceptions: active alcoholism or marijuana).
* In the opinion of the investigator, the participants may have compliance problems with the protocol and the procedures of the protocol.
* Participants with ongoing or recent variceal bleeding (participants can be included 2 weeks after hemorrhagic episode).
* Participants with septic shock at screening.
* Participants with ongoing spontaneous bacterial peritonitis (SBP) infection (participants can be included upon resolution).
* Participants with current infection of coronavirus disease of 2019 (COVID19), those who are less than 14 days post recovery, or those who have clinical signs and symptoms consistent with COVID19 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (66):
- United States (7):
  - Southern California Research Center, Coronado, California
  - University of Miami Hospital, Miami, Florida
  - Rutgers-New Jersey Medical School, Newark, New Jersey
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Missouri Hospital, Columbia, South Carolina
  - Dallas VA Medical Center, Dallas, Texas
  - McGuire VA Medical Center, Richmond, Virginia
- Belgium (3):
  - Université libre de Bruxelles, Brussels
  - Antwerp University Hospital, Edegem
  - UZ Leuven - Campus Gasthuisberg, Leuven
- Bosnia and Herzegovina (3):
  - University Clinical Centre of the Republic Srpska, Clinic for Internal Diseases, Department of gastroenterology, hepatology and toxicology with internal medicine, Mostar
  - Dr. Abdulah Nakas General Hospital, Department of Internal Medicine, Department of Gastroenterohepatology, Sarajevo
  - Zenica Cantonal Hospital, Department of Internal Medicine with hemodialysis, Department of Gastroenterology and hepatology, Zenica
- Bulgaria (8):
  - MHAT "Pazardzhik" Ltd, Pazardzhik
  - MHAT"Sv. Pantelymon", Plovdiv
  - MHAT " Hadzhi Dimitar" Ltd, Sliven
  - MHAT Sliven to MMA Sofia, Sliven
  - MHAT "Sveta Sofia", Sofia
  - UMHAT "Sveti Ivan Rilski", Sofia
  - UMHATEM "N.I.Pirogov", Sofia
  - First Private MHAT Vratsa, Vratsa
- University Health Network - Toronto General Hospital, Toronto, Canada
- Hvidovre University Hospital, Hvidovre, Denmark
- France (5):
  - Hôpital Minjoz - CHU Besaçon, Besançon
  - Hôpital Henri Mondor-Creteil, Créteil
  - CHU de Nice - Hôpital l'Archet 2, Nice
  - CHRU de Strasbourg - Hôpital Hautepierre, Strasbourg
  - Centre Hépato-Biliaire - Hôpital Universitaire Paul Brousse, Villejuif
- Germany (4):
  - Charité - Universitaetsmedizin Berlin, Berlin
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Jena, Jena
- Hungary (5):
  - Magyar Honvédség Egészségügyi Központ Gasztroenterológiai Osztály, Budapest
  - Semmelweis Egyetem I. sz. Sebészeti és Intervenciós Gasztroenterológiai Klinika, Budapest
  - Debreceni Egyetem Klinikai Központ Gasztroenterológiai Klinika, Debrecen
  - Markhot Ferenc Oktatókórház és Rendelőintézet, Eger
  - Albert Schweitzer Kórház, Hatvan
- Italy (3):
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico - S.Orsola, Bologna
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera di Padova, Padua
- Poland (9):
  - Oddział Gastroenterologii i Hepatologii Uniwersyteckie Centrum Kliniczne im. prof.K.Gibińskiego SUM w Katowicach, Katowice
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Zakład Endoskopii SIV 31Aug22, Krakow
  - Oddział Kliniczny Gastroenterologii Ogólnej i Onkologicznej, Uniwersytecki Szpital Kliniczny im. Barlickiego, Lodz
  - Klinika Chorób Wewnętrznych, Diabetologii i Farmakologii Klinicznej, Centralny Szpital Kliniczny, Lodz
  - Oddział Kliniczny Gastroenterologii Ogólnej i Onkologicznej, Uniwersytecki Szpital Kliniczny im. Barlickiego, Lublin
  - ID Clinic, Mysłowice
  - Klinika Gastroenterologii i Hepatologii z Pododdziałem Chorób Wewnętrznych Kliniczny Szpital Wojewodzki nr 1, Rzeszów
  - Centrum Badań Klinicznych, Wroclaw
  - Samodzielny Publiczny Szpital im.Papieza Jana Pawla II, Zamość
- Serbia (9):
  - Clinical Hospital Center "Dr Dragisa Misovic-Dedinje", Clinic for Internal Medicine, Gastroenterology Department, Belgrade
  - Clinical Hospital Center Zvezdara, Clinic for Internal Diseases, Clinical Department for Gastroenterology and Hepatology, Belgrade
  - University Clinical Centre of Serbia, Clinic for Gastroenterology and Hepatology, Belgrade
  - Military Medical Academy, Clinic for Gastroenterology and Hepatology, Belgrade
  - Clinical Hospital Center "Bezanijska Kosa", Clinic for Internal Medicine, Department for Gastroenterology and Hepatology, Belgrade
  - University Clinical Center Kragujevac, Clinic for Internal Medicine, Gastroenterohepatology Center, Kragujevac
  - 'University Clinical Center Nis, Clinic for Gastroenterology and Hepatology, Niš
  - Institution: General Hospital Pančevo, Internal Diseases Department, Gastroenterology Section, Pančevo
  - 'Health Center Uzice, Internal Diseases Department, Gastroenterology Section, Užice
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Universitario Politecnico La Fe, Valencia
- Royal Free NHS Foundation Trust Hospital, London, Londong, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez J, Claria J, Amoros A, Aguilar F, Castro M, Casulleras M, Acevedo J, Duran-Guell M, Nunez L, Costa M, Torres M, Horrillo R, Ruiz-Del-Arbol L, Villanueva C, Prado V, Arteaga M, Trebicka J, Angeli P, Merli M, Alessandria C, Aagaard NK, Soriano G, Durand F, Gerbes A, Gustot T, Welzel TM, Salerno F, Banares R, Vargas V, Albillos A, Silva A, Morales-Ruiz M, Carlos Garcia-Pagan J, Pavesi M, Jalan R, Bernardi M, Moreau R, Paez A, Arroyo V. Effects of Albumin Treatment on Systemic and Portal Hemodynamics and Systemic Inflammation in Patients With Decompensated Cirrhosis. Gastroenterology. 2019 Jul;157(1):149-162. doi: 10.1053/j.gastro.2019.03.021. Epub 2019 Mar 22. PMID 30905652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 410 participants took part in the study at 40 investigative sites across 14 countries in Europe and the United States from 24 July 2018 to 21 May 2024.
Pre-assignment Details: 476 participants with decompensated cirrhosis and ascites were screened of which 410 participants were randomized in a 1:1 ratio to receive either the Standard Medical Treatment (SMT) + Albutein 20% or the SMT alone.
Groups:
- SMT + Albutein 20%: Participants received Albutein 20%, at a dose of 1.5 grams/kilograms (g/kg), based on their body weight (maximum 100 grams per participant), as an intravenous (IV) infusion on Day 1, followed by the same dose of Albutein 20% every 10±2 days along with SMT administered as per institution standards for the management of decompensated cirrhosis up to 12 months.
- SMT Alone: Participants received SMT up to 12 months as per institution standards for the management of decompensated cirrhosis.
Period: Overall Study
Arm/Group | SMT + Albutein 20% | SMT Alone
Started | 203 | 207
Completed | 110 | 105
Not Completed | 93 | 102
Not completed — Death | 44 | 59
Not completed — Withdrawal by Subject | 18 | 13
Not completed — Transplantation | 18 | 12
Not completed — Lost to Follow-up | 4 | 12
Not completed — Physician Decision | 4 | 3
Not completed — Adverse Event | 3 | 3
Not completed — Non-compliance with Study Drug | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized.
Groups:
- SMT + Albutein 20%: Participants received Albutein 20%, at a dose of 1.5 g/kg, based on their body weight (maximum 100 grams per participant), as an IV infusion on Day 1, followed by the same dose of Albutein 20% every 10±2 days along with SMT administered as per institution standards for the management of decompensated cirrhosis up to 12 months.
- Total: Total of all reporting groups
Arm/Group | SMT + Albutein 20% | SMT Alone | Total
Number analyzed (Participants) | 203 | 207 | 410
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (10.03) | 58.7 (10.30) | 58.8 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 55 | 117
  Male | 141 | 152 | 293
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 17 | 35
  Not Hispanic or Latino | 185 | 190 | 375
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 197 | 199 | 396
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Time to Liver Transplantation or Death Through 1 Year After Randomization: Percentage of Participants With an Event
Description: Time to one-year transplant-free survival was calculated as earlier of [(date of liver transplantation or date of death) - randomization date + 1] for participants who died or had liver transplant within the analysis period of 361 days. Participants who neither died nor had liver transplant within analysis period had their time to event censored at earlier of date of last contact or cut-off date. Participants who terminated early for reasons other than death were followed up at months 3, 6, and 12 to collect information on liver transplantation and death, these events if reported by cut-off Day 361, were considered for the endpoint. The percentage of participants with events are presented. The percentage of participants was calculated as [(participants with an event up to the analysis cut-off Day 361) / (number of participants in the ITT group)].
Time Frame: Up to Day 361
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | SMT + Albutein 20% | SMT Alone
Number analyzed (Participants) | 203 | 207
percentage of participants | 33.5 | 38.6
Statistical Analysis 1: Comparison: SMT + Albutein 20% vs SMT Alone; Stratification factors included were the region (Europe or North America) and history of hospitalization for acute decompensation of liver cirrhosis (yes or no); Test type: Superiority; p = 0.17, Cox Proportional- Hazards (PH) model; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.58 to 1.10]

2. Secondary Outcome: Time to Liver Transplantation or Death Through 3 Months After Randomization: Percentage of Participants With an Event
Description: Time to 3-months transplant-free survival was calculated as earlier of [(date of liver transplantation or date of death) - randomization date + 1] for participants who died or had liver transplant within the analysis period of 91 days. Participants who neither died nor had liver transplant within analysis period had their time to event censored at earlier of date of last contact or cut-off date. Participants who terminated early for reasons other than death were followed up at months 3, 6, and 12 to collect information on liver transplantation and death, these events if reported by cut-off Day 91, were considered for the endpoint. The percentage of participants with events are presented. The percentage of participants was calculated as [(participants with an event up to the analysis cut-off Day 91) / (number of participants in the ITT group)].
Time Frame: Up to Day 91
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | SMT + Albutein 20% | SMT Alone
Number analyzed (Participants) | 203 | 207
percentage of participants | 10.8 | 17.9

3. Secondary Outcome: Time to Liver Transplantation or Death Through 6 Months After Randomization: Percentage of Participants With an Event
Description: Time to 6-months transplant-free survival was calculated as earlier of [(date of liver transplantation or date of death) - randomization date + 1] for participants who died or had liver transplant within the analysis period of 181 days. Participants who neither died nor had liver transplant within analysis period had their time to event censored at earlier of date of last contact or cut-off date. Participants who terminated early for reasons other than death were followed up at months 3, 6, and 12 to collect information on liver transplantation and death, these events if reported by cut-off Day 181, were considered for the endpoint. The percentage of participants with events are presented. The percentage of participants was calculated as [(participants with an event up to the analysis cut-off Day 181) / (number of participants in the ITT group)].
Time Frame: Up to Day 181
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | SMT + Albutein 20% | SMT Alone
Number analyzed (Participants) | 203 | 207
percentage of participants | 22.7 | 28.5

4. Secondary Outcome: Time to Death Through 3 Months After Randomization: Percentage of Participants With an Event
Description: Time to 3-months survival was calculated as the earlier of [(date of death) - randomization date + 1] for those participants who died within the analysis period of 91 days. Participants who did not die within the analysis period were censored at the earlier of the date of last contact or analysis cut-off date. Participants who terminated early for reasons other than death were followed up at months 3, 6, and 12 to collect information on death, these events if reported before the analysis cut-off Day 91 of this endpoint, were considered. The percentage of participants with events (death) without censoring participants who underwent liver transplantation within the analysis period were reported. The percentage of participants was calculated as [(participants with an event up to the analysis cut-off Day 91) / (number of participants in the ITT group)].
Time Frame: Up to Day 91
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | SMT + Albutein 20% | SMT Alone
Number analyzed (Participants) | 203 | 207
percentage of participants | 9.4 | 14.0

5. Secondary Outcome: Time to Death Through 6 Months After Randomization: Percentage of Participants With an Event
Description: Time to 6-months survival was calculated as the earlier of [(date of death) - randomization date + 1] for those participants who died within the analysis period of 181 days. Participants who did not die within the analysis period were censored at the earlier of the date of last contact or analysis cut-off date. Participants who terminated early for reasons other than death were followed up at months 3, 6, and 12 to collect information on death, these events if reported before the analysis cut-off Day 181 of this endpoint, were considered. The percentage of participants with events (death) without censoring participants who underwent liver transplantation within the analysis period were reported. The percentage of participants was calculated as [(participants with an event up to the analysis cut-off Day 181) / (number of participants in the ITT group)].
Time Frame: Up to Day 181
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | SMT + Albutein 20% | SMT Alone
Number analyzed (Participants) | 203 | 207
percentage of participants | 16.7 | 23.2

6. Secondary Outcome: Time to Death Through 1 Year After Randomization: Percentage of Participants With an Event
Description: Time to 1 year survival was calculated as the earlier of [(date of death) - randomization date + 1] for those participants who died within the analysis period of 361 days. Participants who did not die within the analysis period were censored at the earlier of the date of last contact or analysis cut-off date. Participants who terminated early for reasons other than death were followed up at months 3, 6, and 12 to collect information on death, these events if reported before the analysis cut-off Day 361 of this endpoint, were considered. The percentage of participants with events (death) without censoring participants who underwent liver transplantation within the analysis period were reported. The percentage of participants was calculated as [(participants with an event up to the analysis cut-off Day 361) / (number of participants in the ITT group)].
Time Frame: Up to Day 361
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | SMT + Albutein 20% | SMT Alone
Number analyzed (Participants) | 203 | 207
percentage of participants | 26.1 | 31.9

7. Secondary Outcome: Total Number of Paracenteses Through 1 Year After Randomization
Description: Paracenteses is a medical procedure used to remove excess fluid from the abdominal cavity. For each participant, the total number of reported paracenteses on treatment was calculated. Number of paracenteses per participant while on treatment was reported.
Time Frame: Up to Day 361
Population: ITT population included all participants who were randomized.
Measure: Mean (Standard Deviation); unit: paracenteses per participant
Arm/Group | SMT + Albutein 20% | SMT Alone
Number analyzed (Participants) | 203 | 207
paracenteses per participant | 1.3 (3.58) | 2.3 (5.07)

8. Secondary Outcome: Number of Participants With Refractory Ascites According to the International Club of Ascites (ICA) Through 1 Year After Randomization
Description: Refractory Ascites was defined as ascites that cannot be mobilized, or the early recurrence of which cannot be prevented because of a lack of response to sodium restriction and diuretic, or the development of diuretic-induced complications that preclude the use of an effective diuretic dosage treatment. Incidence of refractory ascites occurring on treatment was defined as any incidence that occurred with a start date/time on or after the participants date/time of randomization (for SMT Alone group) or commencement of Albutein (SMT+ Albutein 20% group) treatment.
Time Frame: Up to Day 361
Population: ITT population included all participants who were randomized. Overall number of participants analyzed included participants with at least one refractory ascites assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | SMT + Albutein 20% | SMT Alone
Number analyzed (Participants) | 195 | 203
Participants | 33 | 46

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: The Safety population included the subset of participants who received at least one SMT + Albutein 20% administration or SMT alone.
Arm/Group | SMT + Albutein 20% | SMT Alone
All-Cause Mortality (participants affected / at risk) | 53/203 | 67/207
Serious Adverse Events (participants affected / at risk) | 52/203 | 70/207
Other Adverse Events (participants affected / at risk) | 51/203 | 47/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SMT + Albutein 20% (N=203) | SMT Alone (N=207)
Pneumonia (Infections and infestations) | 2 | 8
Urinary Tract Infection (Infections and infestations) | 2 | 7
Sepsis (Infections and infestations) | 2 | 5
COVID-19 Pneumonia (Infections and infestations) | 2 | 1
Septic Shock (Infections and infestations) | 1 | 4
COVID-19 (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 1
Clostridium Difficile Colitis (Infections and infestations) | 1 | 1
Systemic Candida (Infections and infestations) | 1 | 1
Enterococcal Bacteraemia (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Wound Infection (Infections and infestations) | 1 | 0
Clostridium Difficile Infection (Infections and infestations) | 0 | 3
Acute Endocarditis (Infections and infestations) | 0 | 1
Enterococcal Sepsis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Escherichia Sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia Aspiration (Infections and infestations) | 0 | 1
Pneumonia Escherichia (Infections and infestations) | 0 | 1
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal Osteomyelitis (Infections and infestations) | 0 | 1
Staphylococcal Sepsis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Urinary Tract Infection Enterococcal (Infections and infestations) | 0 | 1
Cardiac Failure (Cardiac disorders) | 2 | 1
Cardiac Arrest (Cardiac disorders) | 2 | 0
Cardiac Failure Acute (Cardiac disorders) | 1 | 1
Cardiopulmonary Failure (Cardiac disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Mitral Valve Incompetence (Cardiac disorders) | 1 | 0
Myocardial Injury (Cardiac disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Death (General disorders) | 5 | 4
Sudden death (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Hernia (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 4
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Strangulated incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 3
Seizure (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Coagulopathy (Blood and lymphatic system disorders) | 2 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haematoma (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 3
Renal failure (Renal and urinary disorders) | 0 | 2
Delirium tremens (Psychiatric disorders) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Device dislocation (Product Issues) | 1 | 0
Device breakage (Product Issues) | 0 | 1
Gram stain positive (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SMT + Albutein 20% (N=203) | SMT Alone (N=207)
Hyperkalaemia (Metabolism and nutrition disorders) | 11 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 11
Anaemia (Blood and lymphatic system disorders) | 14 | 17
Urinary tract infection (Infections and infestations) | 13 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 2
Diarrhoea (Gastrointestinal disorders) | 11 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor 30 days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to 120 days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT03451292/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT03451292/SAP_001.pdf